CLINICAL TRIAL: NCT01852682
Title: A Phase III Study of PA21 in Peritoneal Dialysis Patients With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA1303
Record Dates: First submitted 2013-05-07; First posted 2013-05-14 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Peritoneal Dialysis; Hyperphosphatemia
Keywords: Peritoneal Dialysis; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

ARMS (1):
- PA21 (Experimental)
  Interventions: Drug: PA21

INTERVENTIONS:
Drug: PA21

SUMMARY:
The purpose of this study is to investigate efficacy and safety, when administering PA21, in peritoneal dialysis patients having hyperphosphatemia.

ELIGIBILITY:
Inclusion Criteria:

* Receiving stable maintenance peritoneal dialysis
* Peritoneal dialysis patients with hyperphosphatemia

Exclusion Criteria:

* Patients having history of a pronounced brain / cardiovascular disorder
* Patients having severe gastrointestinal disorders
* Patients having severe hepatic disorders

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Serum phosphate concentrations | 12 weeks

SECONDARY OUTCOMES:
Incidences of Adverse Events | 12 weeks
Incidences of Adverse Events | 28 weeks
Serum phosphate concentrations | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo and Other Japanese City, Japan